A randomized controlled trial to assess the performance and safety of a novel Ostomy Ring (Osto Ring<sup>™</sup>) to improve ileostomy and colostomy management Eugene Yen, MD, K. Agnes Brugger BSN, RN

### **Background and Significance:**

Ostomy surgery refers to a surgical procedure in which part of the intestine is removed and the intestinal contents are rerouted through the abdominal wall via a stoma (<a href="http://www.niddk.nih.gov/health-information/health-topics/digestive-diseases/ostomy-surgery-bowel/Pages/ez.aspx">http://www.niddk.nih.gov/health-information/health-topics/digestive-diseases/ostomy-surgery-bowel/Pages/ez.aspx</a>). This type of surgery results in the patients utilizing an external pouch, a plastic bag affixed around the stoma on the abdominal skin to collect the waste. Depending on the reason for the surgery, stomas may be temporary or permanent.

It was estimated in 2012 that there are 1 million people in the United States and Canada living with ostomies, with an additional 100,000 new ostomies created per year in the United States. (Mitchell KA, Rawl SM, Schmidt CM, et al. Demographic, clinical, and quality of life variables related to embarrassment in veterans living with an intestinal stoma. J Wound Ostomy Continence Nurs. 2007;34(5):524-532).

The quality of life for patients who undergo this type of surgery is significantly affected. It is an adjustment for a patient to psychologically understand that his or her body will no longer perform a bodily function "normally". The patient needs to learn new skills such as how to correctly apply the pouching system, adjust wear time, and learn how and when to empty the pouch and remember to check the pouch seal to detect any signs of leakage. These new skills take time to learn and one of the greatest challenges is to find the best pouching system that can provide a consistent wear time to prevent leakage, embarrassment and peristomal skin issues.

A new device has been created with the aim of improving wear time and decreasing problems with leakage. The Osto Ring<sup>™</sup> (GoDuRn LLC, 9722 Oak Pass Rd., Beverly Hills, CA 90210) is a novel and proprietary add-on modifier to the Hollister 2 piece New Image pouching system that creates a more secure seal between the patient's peristomal skin and the skin barrier, and therefore reduces the risk of leakage.

We hypothesize that the addition of the Osto-Ring<sup>™</sup> will reduce leakage from the stoma appliance and may also increase the length of time needed between pouch changes. Currently, the mean ostomy pouch wear time in the United States is 5.2 days (Richbourg L, Fellows J, Arroyave WD. Ostomy pouch wear time in the United States. J Wound Ostomy Continence Nurs. 2008 Sep-Oct;35(5):504-8), and out-of-pocket costs can be as high as \$30 with each pouching system change which translates to a yearly cost of close to \$3000. Longer wear time would therefore translate into needing fewer ostomy bags and less money spent on ostomy supplies.

#### **Overall Objective:**

The primary objective of this pre-market study is to assess the safety and performance of the Osto  $Ring^{TM}$  as it relates to the pouching system wear time and degree of leakage.

#### **Research Design:**

Study population: 30 adult subjects who have had an ileostomy or colostomy for at least 6 months, who currently use the Hollister New Image 2 piece pouching system acting as their own controls, will use their standard 2 piece New Image Hollister pouching system without the Osto Ring<sup>™</sup> for 28 days. On Day 29 subjects will be switched to the Osto-Ring regimen until day 56. Patients will be evaluated in person at Day 0 and approximately Days 28, 56, and 75 (within business days and scheduling convenience).

The Osto-Ring for this study is being supplied by GoDuRn, LCC, and provided to subjects free of charge.

During the standard of care visit to the health care provider, subjects will be evaluated to confirm that they meet the criteria for participating in this study.

#### Study Design:

#### Day 0-27

#### **Visit One**

- Subject will wear their standard of care Hollister 2 piece New Image pouching system for 28 days.
  - At the first visit they will remove their pouching system to allow the investigator to assess their skin (research staff will take photo) using the Ostomy Skin Tool Reference Guide [See appendix B]
  - They will be given and asked to fill out the Quality of Life Questionnaire [See appendix C]
  - They will be given Ostomy Evaluation Record [See appendix A] and asked to complete this at every pouching system change. (And take photos of the skin site and adhesive side of the ostomy flange.)

#### Day 28-55

#### **Visit Two**

- Subjects will now wear their standard of care Hollister 2 piece New Image pouching system with the Osto-Ring for the next 28 days.
  - At the first visit they will remove their pouching system to allow the investigator to assess their skin using the Ostomy Skin Tool Reference Guide [see appendix B] (photo taken)
  - They will be fitted for the proper Osto-Ring size and given a belt.
  - They will be given and asked to fill out the Quality of Life Questionnaire [See appendix C]
  - They will be given 2 questionnaires and asked to complete them at every pouching system change. Subject will take photograph at each stoma change
    - Ostomy Evaluation Record [See appendix A]
    - Osto Ring Evaluation Record [See appendix D]

#### **Day 56**

#### Visit Three

Patients will decide if they want to continue using the Osto-Ring<sup>™</sup> with their standard of care pouching system.

 Their pouching system will be removed and will have a skin assessment by the investigator using the Ostomy Skin Tool Reference Guide, Appendix B.

- They will be asked how they are doing and to report any side effects they may have experienced even if they do not think it is related to the Osto-Ring<sup>TM</sup>.
- They will be asked to complete :
  - The Ostomy Quality of Life Questionnaire

If they felt that the Osto Ring was helpful, subjects will be asked to extend the wear of their devices by 1-4 days per their experience (if possible). Photographs will be taken at each stoma change of the skin and the adhesive side of the flange.

#### **Day 75**

#### **Visit Four**

At this last visit, patients can decide to have their Osto Ring removed or continue using it if they like.

All four of the clinic visits are considered research-related, along with completion of questionnaires and peristomal skin assessment.

During this study, Dr. Yen and his research team will collect information about the patients for the purposes of this research. This includes their name, telephone number, medical record number, initials, date of birth, medical, surgical and medication history, date of study entry, dates of study procedures and results of tests and procedures done as part of the study.

To calculate the study sample size, data from prior studies and expert opinion was used for power analysis since this device uses a novel approach to increase wear time. The mean wear time for ileostomy pouches in the United States is 5.01 +/- 2.25 days (Richbourg L, Fellows J, Arroyave WD. Ostomy pouch wear time in the United States. J Wound Ostomy Continence Nurs. 2008 Sep-Oct;35(5):504-8). An increase of wear time by 25% to 6.26 days is beneficial for patient care. We determined the effect size to be 0.56 assuming that the pool standard deviation is similar to the study cited above. Using a paired t-test with a significance level of 0.05 and power of 0.8, 27 patients are needed for this study.

All patients will be recruited from the NorthShore University HealthSystem IBD center and General Surgery Clinics. Evaluation and management for any stoma related questions, concerns or assessments may also be provided by our IBD center team. Results of the study will not be made available to the sponsor or anyone with a perceived or actual conflict of interest (eg actual/potential financial relationship) until the statistical analysis has been independently completed.

#### **Inclusion Criteria:**

Subjects interested in participating in the clinical investigation must comply with the following criteria:

- 1. Are at least 18 years of age and have full legal capacity
- 2. Have had an end or loop ileostomy or colostomy for at least 6 months.
- 3. Have used a Hollister 2 piece New Image pouching system for at least 8 weeks
- 4. Able to provide informed consent
- 5. Have a stoma with a diameter of 57mm or less

6. Change their pouching system at least two times in seven days

#### **Exclusion Criteria:**

Subjects complying with the following criteria must be excluded from participation in the clinical investigation:

- 1. Unable to give informed consent.
- 2. Are pregnant or currently breastfeeding.
- 3. In the last 2 months has received or is currently receiving, chemotherapy or radiation therapy.
- 4. In the last month has received or is currently receiving systemic or local steroid treatment in the peristomal area.
- 5. Currently suffering from severe peristomal skin problems such as peristomal pyoderma, abscess.
- 6. Currently suffering from a peristomal hernia.
- 7. Known hypersensitivity toward any of the test product (Osto Ring<sup>™</sup> is made of surgical grade stainless steel)
- 8. In the last 30 days has participated or is currently participating in a clinical study
- 9. Assessed with an ostomy skin tool score of ≥3

#### **Primary Outcomes:**

#### <u>Performance Efficacy</u>:

To evaluate the Osto  $Ring^{TM}$  for pouching system wear time, and degree of leakage in subjects when using the Osto  $Ring^{TM}$  as compared to when not using the Osto- $Ring^{TM}$ 

- Integrity of the adhesive side of the flange (photos)
- Wear Time:
  - Total time pouching system worn will be calculated by the Ostomy Evaluation Record.
     This is defined as the difference between the dates and times the appliance is changed.
     (Appendix A)
- Leakage:
  - Degree of leakage at time of pouching system changes will be measured using line item from Ostomy Evaluation Record (Appendix A)

#### **Secondary Outcomes:**

- 1. The condition of the peristomal skin and stoma (Appendix B)
- 2. The number and frequency of adverse events
- 3. The subjects' quality of life using the Stoma Quality of Life (QoL) questionnaire (Appendix C)
- 4. Subject Ease of Use (ease of application, pain level with application, comfort, convenience of use) will be assessed using Likert scale: 1 = poor, 2 = satisfactory 3= very good, 4= excellent (Appendix D)

#### **Analysis plan:**

All means and frequencies will be compared between the groups with the Osto Ring<sup>TM</sup> versus the group without it and will be controlled for the order in which a subject used the Osto Ring.

#### • Wear Time:

o Mean days in between pouching system changes

#### <u>Leakage:</u>

- o Frequency of any degree of leakage at pouching system changes
- o Frequency of much leakage at time of pouching system change

#### • Skin condition:

- o % of patients with moderate to severe skin conditions at time of each WOC nurse or physician study visit
- o Mean % of time with moderate to severe skin conditions throughout the 4 week interval at every WOC nurse or physician study visit

#### Quality of Life:

o Mean quality of life scores

#### • Time per Ostomy Care Session

o Mean minutes spent during ostomy care session

#### • Ease of Use

- Mean % of time ease of use reported as very good or excellent by subject , <u>Satisfaction and Confidence</u>
  - o Mean satisfaction and confidence scores
- Device Recommendation
- o % of subjects reporting they strongly agree to recommend the device to others We will compare the baseline characteristics of the two groups. Continuous variables will be compared with the paired *t* test, and categorical variables were compared with the Fisher exact test. Each item on the ostomy evaluation record form will be individually reported.

#### Safety Assessments and Termination Guidelines

WOC nurses will perform skin assessments at key times. Patients are to be told that they must mention any deviation from their baseline ostomy pouching system changing routine. Failure to do so will result in a protocol violation. Patients receiving an Ostomy Skin Tool score of ≥3 without a known cause will be withdrawn from the study.

Any patient suffering an allergic reaction to either product (the standards New Image Hollister appliance or Osto Ring) or suspected of having an adverse reaction of any kind as determined by the patient and/or the ostomy will be removed from the trial, return for clinical assessment as indicated and return to their standard stoma care appliance.

The data safety monitoring committee will consist of Drs Eugene Yen and Joseph Muldoon, who will review any unanticipated adverse events and have the authority to stop the trial at any time if any safety concerns are raised.

### Osto-Ring<sup>TM</sup> Risks

Side effects may include:

- allergic reaction to the ring,
- worsening of the peristomal skin condition, or
- prolonged time needed in changing the ostomy pouching device.

### **2-piece New Image Hollister Pouching System**

The 2 piece New Image Hollister Pouching System is standard of care. Concerns regarding this system will be handled by the regular physician. However, all concerns will be addressed.

Appendix A

Dated 4/22/19

# **OSTOMY EVALUATION RECORD**

| ID Number:<br>Number of days since | Da<br>e last Change: | ate: |
|---|---|---|
| - | • • | ing items describing your experience in between pouching<br>luation Record should accompany EACH Ostomy Change |
| 1. What was | • | me (time between placing the pouching system on and taking |
| 2. Did you n | otice any skin damage | e around your stoma, redness and open areas? Yes or No |
| □ No odor<br>(Skip to Ques<br>4. How both | stion 3)<br>ersome did you consid | ostomy between appliance changes? Slight odor Strong odor der the odor? |
| □ Not at all b | | |

| | ☐Slightly bothersome<br>☐Moderately bothersome<br>☐Severely bothersome | | |
|---|---|---|---|
| | Extremely bothersome | | |
| 5 | . Did you encounter leakage and if | so how much? | |
| (9 | □No leakage<br>Skip to Question 7)<br>ow many days was the pouching sy | □Slight leakage<br>□Much leakage<br>stem in place befor | e you noted leakage? |
| 6 | . How bothersome did you consider | the leakage? | |
| | □Not at all bothersome □Slightly bothersome □Moderately bothersome | | ☐ Severely bothersome ☐ Extremely bothersome |
| 7 | . Was your social freedom limited b | y your ostomy? | |
| | Not limited at all | ☐ Slightly limited | ☐Greatly limited ☐Very unaccepting |
| | omewhat unaccepting | _ | |
| | . How convenient was your ostomy | care? | |
| | □Very convenient<br>□Somewhat convenient | | 8. How satisfied were you with your |
| | ]Neutral | | ostomy care? |
| | ∃Somewhat inconvenient<br>∃Very inconvenient | | □ Very satisfied □ Somewhat satisfied □ Neutral □ Somewhat dissatisfied □ Very dissatisfied □ Somewhat dissatisfied □ Very dissatisfied □ Very dissatisfied |
| severity o<br>(DET). (M | my Skin Tool is a standardized and v<br>f peristomal skin change in terms of | discoloration (D), 6 | g instrument for assessing the extent and<br>erosion (E), and tissue overgrowth (T)<br>0, 932-4) Ostomy Skin Tool used with |
| Date: | Subject ID | | |
| If area | iscoloration (1-3) | | |

| Severity of Discoloration (1-2) | |
|---|---|
| Erosion Area of Erosion (1-3) If area is 0 then severity must be 0 | |
| Severity of Erosion (1-2) | |
| Tissue Overgrowth Area of tissue overgrowth (1-3) If area is 0 then severity must be 0 Severity of tissue overgrowth (1-2) | |
| Total OSTOMY SKIN TOOL REFERENC | E GUIDE |



Ostomy Skin Tool used with written permission from Coloplast, Minneapolis, MN.

## Appendix C

Ostomy Quality of Life Questionnaire

| 1. | I feel the need to know where the nearest toilet is | | | |
|---|---|---|---|---|
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |
| 2. | l become anxiou | us when the pouch is full | | |
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |
| 3. | I feel tired durin | g the day | | |
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |
| 4. | I am afraid of m | eeting new people | | |
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |
| 5. | It is difficult to h | nide the fact that I wear a pouc | h | |
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |
| 6. | My stoma make | s it difficult for me to be with o | other people | |
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |
| 7. | I sleep badly du | ring the night | | |
| | Always | Sometimes | Rarely | Not At All |
| | 1 | 2 | 3 | 4 |

8. I feel lonely even when I am with other people

| Always | Sometimes Rare | | Not At All |
|---|---|---|---|
| 1 | 2 | 3 | 4 |
| 9. I need to rest duri | ng the day | | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 10. I worry that my co | ondition is a burden to peopl | e close to me | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 11. I avoid close phys | ical contact with my friends | | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 12. I worry that my fa | mily feel awkward around n | ne | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 13. I feel embarrassed | d about my body because of | my stoma | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 14. It would be difficu | ılt for me to stay away from | home overnight | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 15. I worry that the p | ouch rustles | | |
| Always | Sometimes | Rarely | Not At All |
| 1) | (2) | (3) | <b>(4)</b> |

| 16. I worry that the po | ouch may smell | | |
|---|---|---|---|
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 17. My stoma makes | me feel sexually unattractive | <b>e</b> | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 18. I worry about nois | ses from the stoma | | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 19. I worry that the po | ouch will loosen | | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |
| 20. My stoma pouch l | imits the choice of clothes th | nat I can wear | |
| Always | Sometimes | Rarely | Not At All |
| 1 | 2 | 3 | 4 |

## Appendix D

| 1. | Osto-Ring <sup>TM</sup> | <b>Evaluation</b> | Record |
|----|-------------------------|-------------------|--------|
|----|-------------------------|-------------------|--------|

| | very<br>easy<br>5 | somewhat<br>easy<br>4 | neutral<br>3 | somewhat<br>difficult<br>2 | very<br>difficult<br>1 |
|---|---|---|---|---|---|
| 2. | Satisfacti | on with Osto Ring <sup>™</sup> | | | |
| | Poor | Satisfacto | ory | Very Good | Excellent |
| | 1 | 2 | | 3 | 4 |
| 3. | Confiden | ce with Osto Ring™ | | | |
| | Poo | or Satisf | actory | Very Good | Excellent |
| | 1 | (2 | ) | 3 | 4 |
| 4. | Problems | s with Osto Ring <sup>TM</sup> | | | |
| | No | ne Few | | Several | Many |
| | 1 | 2 | ) | 3 | 4 |
| Ple | ase specify ar | ny problems: | | | |
| 5. | Comfo | ort of Osto Ring™felt | | | |

| very | somewhat | neutral | somewhat | very |
|-------------|-------------|---------|---------------|---------------|
| comfortable | comfortable | | uncomfortable | uncomfortable |
| 5 | 4 | 3 | 2 | 1 |

I would highly recommend the Osto  $\mathsf{Ring}^\mathsf{TM}$  to others

| | Strongly Agree | Agree | Neither | Disagree | Strongly Disagree |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | (\$) |
| 6. | Have you chan | iged your pouch | iing system in any way | ? | |
| | | Yes | | No | |
| 7. | Is there any | thing else that y | you would like to tell u | s about the Osto | Ring <sup>™</sup> device? |